CLINICAL TRIAL: NCT00331942
Title: Study of Breast Cancer Associated Antibodies
Brief Title: Breast Cancer Associated Antibodies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lab Discoveries Ltd. (Industry)
Other Study IDs: LD-BC-CAAb
Record Dates: First submitted 2006-05-27; First posted 2006-05-31 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2006-04

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Associated; Antibodies
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To determine the ability of the Cimmunology process to lead to in vitro antibody production, the ability of the ELISA assays to detect any of those antibodies, and to establish the relationship between the ELISA results and the clinical / pathological status of the patient. The statistical significance of the CAAb test results will be determined.

DETAILED DESCRIPTION:
General Information

Antibodies are a specific response to any "foreign" antigen, and they are usually detectable in the serum within 5-7 days after the initial exposure to it. However, there are some cases where there is a suppression of the specific immune response, such as in the case of a tumor. To date, there are no reports on serum antibodies that are associated to cancer. Some tumors, when surgically removed and studied have been found to have both infiltrates of T lymphocytes and antibodies bound to the tumor cells. These antibodies (and other specific immune responses) are assumed to be formed at later stages of the tumor growth, however, even in those cases, serum antibodies have not been reported (probably due to them being mostly "absorbed" by the tumor mass).

Since the mutations of a normal cell that lead to a malignant cell mass involves changes in the structure and function of the cells, it could be assumed that the immune system has recognized some of these changes as antigenic determinates that should be responded against; if so, than the suppression caused by the tumor would be the reason for the lack of antibodies.

If this immune suppression could be overcome, in vitro, it could lead to the formation of antibodies that are not detectable in the serum (We call this process Cimmunology). Identifying the structures that the antibodies bind to, and looking for a correlation between the tumor pathology and the antibodies' specificity - could provide additional information about the tumor - via a blood test.

1.2 Future CAAb Test

The Cimmunology based test is comprised of an in-vitro stimulation step and an antibody detection step.

The assay will be used to find cancer associated antibodies in Breast cancer patients.

Identification of Breast cancer associated antibodies could provide the clinician with additional immunological and antigenic information regarding the patient's condition or medical status.

The Cimmunology process is comprised of a blood collection and processing step and an incubation (in a special stimulation "tube" called CimTube) period in a humid, 37oC incubator with 5% CO2.

The test for the detection of specific antibodies is ELISA based, and includes different potentially interesting antigens.

The relevant medical and pathological information, to be collected form the patient's file, will enable a more detailed analysis of the test results.

0 STUDY OBJECTIVES

2.1 Primary objective

To find Cancer Associated Antibodies

2.2 Effectiveness

To determine the ability of the Cimmunology process to lead to in vitro antibody production, the ability of the ELISA assays to detect any of those antibodies, and to establish the relationship between the ELISA results and the clinical / pathological status of the patient. The statistical significance of the CAAb test results will be determined.

3.0 STUDY POPULATIONS AND PATIENT SELECTION

3.1 Study Population

3.1.1 Breast cancer patients The study population will include subjects that have been diagnosed with suspected breast cancer, i.e. positive biopsy, prior to any surgical procedure (or any other anti-cancer treatment).

3.1.2 Control group

The control group will include patients, at breast cancer centers or any other appropriate care unit, with negative Mammography in the last 3 months.

3.2 Participating Centers

3.2.1 General - The study will be based on multi-centers participation.

3.2.2 Locations - All sites will be within Hospitals, either in the Breast Cancer centers or in the relevant specific unit which is responsible for providing care for the BC patients. The minimum number of sites for the study is 2 and the max is 10.

STUDY DESIGN

4.1 Overall Description

The current study is a comparative observational two-arm study, involving all consecutive Breast cancer patients during the study duration, and age matched control subjects. The purpose of the study is to assess the effectiveness of the CAAb test in detecting Breast cancer associated antibodies.

Subjects will be screened for potential participation in the study, according to the inclusion and exclusion criteria. Patients recruited will be asked to sign an informed consent form.

The data on the patients will include parameters of the clinical and pathological state of the patients, results of CimTube culture step and the experimental kits. The effectiveness of the CAAb test will be assessed by evaluating the statistical significance of the CAAb test used.

The study will utilize a three step group-sequential design with two interim and one final analysis using the O'Brian-Fleming' boundaries. The data collection may be stopped after the first or second interim analysis if the bounds are reached. This could substantially decrease the number of patients and the time of the study, while just slightly increasing the maximum number of patients. (See Sample size considerations below).

We will use 1:2 ratio between cancer and control patients to decrease the necessary number of cancer patients which is the main limiting factor.

The sponsor will conduct interim analysis, following the first third and second third of Breast cancer cases and the sample size will be recalculated accordingly to the obtained estimates of the mean and variance of the test in the two groups.

Therefore, at least 100 patients will be enrolled in the study. The control group will be of 200 patients.

4.2 Study Procedure

In the hospital,

First, an identified study patient has to sign an informed consent form, and her Eligibility Form filled (see appendix B), both should be bar-coded.

Patient demographic and clinical information acquired from the patient's medical file, including age, country of origin, medical history and results of tests done leading to the diagnostic evaluation of Breast cancer (not relevant in the control group) will be recorded on the appropriate, bar-coded, pre-study case report forms (see appendix C, CRF-BC and CRF-BC-Control). The reports will be either electronic (a dedicated and secured internet site) or via a hard copy. A hard copy of the records will be kept in the department. The study is anonymous and the Department will keep the name of the patient without reveling it to investigators and to the study sponsor.

The Study Sponsor will provide the tubes and the barcode labels for monitoring. The doctor/ nurse/ phlebotomist will collect three heparin vacuum tubes (20-24 ml), label (bar-code) them, and fill up the initial step in the "Sample follow-up form" (SFF) (see appendix D). The tubes with the blood will be packaged in double sealed containers (will be provided by the sponsor). The department will notify the designated shipper to collect the blood up to 1 hour from the time that it has been sampled.

For each BC sample two age matched controls (+/- 3 years) will be recruited too.

Transportation from the Hospital to the Handling Lab

The blood will be transported at room temperature (18-250C), according to the relevant regulations, to the laboratory. Transportation time will be not more than 6 hours. Times to be recorded in SFF.

In the blood handling laboratory:

The blood handling laboratory (to be located no further than 200km from the collection site) will isolate PBMC (Peripheral blood mononuclear cells) and put them into Cimmunology culture within 20 hours form the sampling time (fill up time in SFF).

The detailed protocol and the Cimmunology media will be provided by Lab Discoveries to the participating laboratories (where applicable). All hospitals in Israel will send the blood samples to the laboratory at Lab Discoveries. After the culture step, the culture fluid will be collected and frozen at -80, in properly labeled aliquots. The frozen samples will be sent to the diagnostic laboratory for antibody tests.

In the diagnostic laboratory:

Antibody tests, such as ELISA, will be prepared using different antigens. The samples will be tested for response to the two antigens that have been identified in the past, and for additional new ones. All the data will be permanently recorded directly into a dedicated computer. For each sample all antibody results will be put into the coded patient file. The results will be analyzed by a statistician with expertise in cancer population studies.

At the Hospital, post surgery:

2-3 weeks after the surgery, the CRO will collect from the patient's file the results from the pathology lab and any other relevant information as to the nature and state of the tumor that was removed during surgery. These results will be recorded on the dedicated and secured internet site and a printed bar-coded CRFs will be kept in the Department.

9.0 STATISTICAL CONSIDERATIONS

The present study is a comparative observational two-arm study, involving all consecutive Breast cancer patients during the study duration, and age matched control subjects. The main purpose of the study is to assess the effectiveness of the CAAb tests. This effectiveness will be measured by the Fisher' distance (often called "effect size") d defined as

Where m1 is the mean value of the test in the controls, m2 is the mean value in the Breast cancer patients, |m1-m2| denotes the absolute value of the difference (m1-m2), and s is the common estimate of the standard deviation of the distribution of the test in one group (control or Breast cancer).

9.1 Statistical Hypothesis

Null Hypothesis: There is no relationship between the presence or absence of BC and the CAAb i.e. d=0

Alternative hypothesis: The expectation of the CAAb in the cancer population differ from that of the control population…. i.e. m1 not equal to m2 Since the sign of the difference is not important the test will be two-sided.

9.2 General Considerations

According to our previous results, we assume that

1. The distributions of the test results in each group are close to Normal or may be transformed to the Normal by log-transformation.
2. The variance of the distributions in the two groups are approximately equal
3. Having in mind that this is a pilot study we will consider the results as significant if the two-sided p-value is 0.1 or less. The bound 0.1 instead of 0.05 was chosen to decrease the chances of random exclusion of some potentially informative tests.

When deciding the continuation of the study no correction for multiple comparisons is assumed. However, the results will be presented without and with the correction using the FDR of Benjamini&Hochberg approach (Benjamini, Hochberg 1995).

Where confidence limits are appropriate, the confidence level will be 95% .

9.3 Sample Size The sample size was calculated using relevant information from our previous study on Peptides P3 and P1 and Breast cancer. There is no information in the literature regarding cancer associated antibodies.

The sample size is calculated for a three step sequential group design with two sided significance 0.1 and 0.05, power 0.8, for cancer : control ratio 1:2, for D of 0.5. The calculations used the standard formulas for sample size necessary for comparison mean values in two independent groups by t-test. The correction for a group-sequential procedure with O'Bien and Fleming's test increases the numbers by 1.017 and 1.027 for significance values 0.05 and 0.1, that is negligible for our sample sizes. (see C. Jennison, B.W.Turnbill Group Sequential Methods with Applications to Clinical Trials Chapmann&Hall(2000) Boca Raton FL US pp30 table 2.4).

The calculations were done using NCSS-PASS software.

9.4 Endpoints Evaluation

9.4.1 Effectiveness Analysis

A calculated D between 0.3 and 0.5 will mark a test as non effective to be used alone. However, it may be important in combination with other tests as a part of the multivariate test procedure. Tests with d<0.3 will be considered as non-effective. A test, or a combination of tests, with d>0.5 will mark the CAAb test as effective.

ELIGIBILITY:
Inclusion Criteria BC:

* Subjects 18 years or over.
* Patients diagnosed with suspected breast cancer, (positive mammography or ultrasound or physical examination) and have a positive biopsy.
* Patients willing to participate as evidenced by signing the written informed consent.

Exclusion Criteria BC:

* Subjects less than 18 years
* Patients with prior history of other tumors (except skin cancer)
* Hematologic systemic disorders
* Patients that have undergone chemotherapy
* Patients that have been under anesthesia in the last three months.
* Patient not willing to sign written informed consent.

Inclusion Criteria Control -

* Subjects 18 years or over
* Patients willing to participate as evidenced by signing the written informed consent
* Subjects had a negative mammography in the past three months.

Exclusion Criteria Control -

* Subjects less than 18 years
* Hematological malignancies
* History of any past tumors
* Other breast pathology
* Patients that have been under anesthesia in the last three months
* Patients treated with immuno-suppressant drugs
* Patient not willing to sign written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-07; Study Completion 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Tamar J Cohen, Phd., Principal Investigator — Lab Discoveries
Locations (2):
- Israel (2):
  - Soroka, Beersheba
  - Carmel Medical center, Haifa